CLINICAL TRIAL: NCT05261464
Title: Heart Rate Controller in Computed Tomography Coronary Angiography: A Randomized Controlled Trial of Metoprolol, Diltiazem and Ivabradine
Brief Title: Heart Rate Controller in Computed Tomography Coronary Angiography
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Si047/2021
Record Dates: First submitted 2022-02-06; First posted 2022-03-02 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Heart Rate; Coronary Computed Tomography Angiography
Keywords: coronary computed tomography angiography (CCTA); Target Heart rate
MeSH Terms: interventions — Metoprolol; Ivabradine; Diltiazem

STUDY DESIGN:
Intervention Model Description: 1. Extract patients who undergo routine Computed Tomography Coronary Angiography (CCTA) with heart rate (HR) > 60 bpm at rest
  2. Enroll patients using Inform consent from the first date of study period until reach the required sample size
  3. Randomize patients to 1:1:1 using 6 block randomization by nQuery program
  4. Assign sequential encapsulated drugs distribute from Siriraj's dispensary to patients according to randomization and protocol prior to CCTA.
  5. Assigned encapsulated until patient reaches target HR or until full dose according to each drugs protocol prior to CCTA.
  6. Continuous monitor blood pressure and heart rate every 15 minutes and closed observe side effects and complication until at least 1 hr after finish CCTA.
  7. Review medical record and CCTA results, then fill in case record forms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: We blinded both investigators and patients using encapsulated drugs distribute from Siriraj's dispensary and randomly assign to our patients. These encapsulated drugs then were sealed from humidity and kept at temperature below 25 degree celsius . These drugs will not be kept for more than 1 week after encapsulated. These encapsulated were assigned according to serial number generate from nQuery program by pharmacist Siriraj's dispensary. In each package, the number from first to fourth encapsulated drugs were assigned from Siriraj's dispensary in order to prescribe to patient when HR can not reach target prior to CCTA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Metoprolol protocol (Active Comparator): 1. Metoprolol tartrate 50 mg will be given if patient's HR is more than 60 bpm.
  2. Monitor BP and heart rate HR every 15 minute to assess targeted HR and side effects until patient's is sent to CCTA.
  3. If patient can not reach targeted HR (less than 60 bpm) at 30 minutes, then second dose of 50-mg metoprolol will be given.
  4. If patient can not reach targeted HR at next 30 minutes, then third dose of 50-mg metoprolol will be given.
  5. If patient can not reach targeted HR at next 30 minutes, then fourth dose of 50-mg metoprolol will be given.
  6. If patient's HR reach targeted HR for 15 minutes apart for 2 times or received total dose of 200 mg metoprolol tartrate, then total time will be recorded and patient will proceed to CCTA.
  7. If patient can not reach targeted HR according to protocol, cardiac imaging specialist will decide whether to give further medication for HR control or proceed to CCTA. Cardiac imaging specialist may be able to consult dispensary.
  Interventions: Drug: Metoprolol tartrate
- Ivabradine protocol (Experimental): 1. Ivabradine 5 mg will be given if patient's HR is more than 60 bpm.
  2. Monitor BP and heart rate HR every 15 minute to assess targeted HR and side effects until patient's is sent to CCTA.
  3. If patient can not reach targeted HR (less than 60 bpm) at 30 minutes, then second dose of 5-mg Ivabradine will be given.
  4. If patient can not reach targeted HR at next 30 minutes, then third dose of 5-mg Ivabradine will be given.
  5. If patient can not reach targeted HR at next 30 minutes, then placebo will be given.
  6. If patient's HR reach targeted HR for 15 minutes apart for 2 times or received total dose of 15 mg ivabradine with 1 dose of placebo, then total time will be recorded and patient will proceed to CCTA.
  7. If patient can not reach targeted HR according to protocol, cardiac imaging specialist will decide whether to give further medication for HR control or proceed to CCTA. Cardiac imaging specialist may be able to consult dispensary.
  Interventions: Drug: Ivabradine
- Diltiazem protocol (Experimental): 1. Diltiazem immediate release (IR) 30 mg will be given if patient's HR is more than 60 bpm.
  2. Monitor BP and heart rate HR every 15 minute to assess targeted HR and side effects until patient's is sent to CCTA.
  3. If patient can not reach targeted HR (less than 60 bpm) at 30 minutes, then second dose of 30-mg diltiazem will be given.
  4. If patient can not reach targeted HR at next 30 minutes, then third dose of 30-mg diltiazem will be given.
  5. If patient can not reach targeted HR at next 30 minutes, then fourth dose of 30-mg diltiazem will be given.
  6. If patient's HR reach targeted HR for 15 minutes apart for 2 times or received total dose of 120 mg 30-mg diltiazem IR, then total time will be recorded and patient will proceed to CCTA.
  7. If patient can not reach targeted HR according to protocol, cardiac imaging specialist will decide whether to give further medication for HR control or proceed to CCTA. Cardiac imaging specialist may be able to consult dispensary.
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Drug: Metoprolol tartrate — Prescribe oral metoprolol tartrate according to doses and time duration until patient reach targeted HR of less than 60 bpm or maximize dose according to each drug protocols prior to CCTA.
  Arms: Metoprolol protocol
Drug: Ivabradine — Prescribe oral ivabradine according to doses and time duration until patient reach targeted HR of less than 60 bpm or maximize dose according to each drug protocols prior to CCTA.
  Arms: Ivabradine protocol
Drug: Diltiazem — Prescribe oral diltiazem immediate-release according to doses and time duration until patient reach targeted HR of less than 60 bpm or maximize dose according to each drug protocols prior to CCTA.
  Arms: Diltiazem protocol

SUMMARY:
Coronary computed tomography angiography (CCTA) is one of important non-invasive test for diagnosis of coronary artery disease. Cardiac motion artifact by heart rate (HR) has impact on CCTA interpretation. Current recommendation suggests HR reduction at less than 60 bpm with using of oral metoprolol. However, there are populations that are contraindicated for beta blockers. There were scantly data of calcium channel blocker and ivabradine. Moreover, there is no data comparing these 3 drug groups within single trial This double-blinded randomized controlled trial compares oral metoprolol immediate release, diltiazem immediate release and ivabradine with primary endpoint of patients' percentage to achieve target HR lower than 60 bpm prior to CCTA.

DETAILED DESCRIPTION:
Coronary computed tomography angiography (CCTA) is one of important non-invasive test for diagnosis coronary artery disease. Information of CCTA can provide information such as coronary artery lumen, vessel wall, degree of stenosis and component of coronary arterial plaque. Most of studies in CCTA represent high negative predictive value (NPV) approximately 93-100 %.However, motion artifact has impact on CCTA interpretation, especially when heart rate (HR) at more than 70 beat-per-minute (bpm). Therefore, HR reduction maneuver is necessary for CCTA. Current recommendation suggests HR reduction at < 60 bpm for best quality of CCTA imaging and to minimized duration of exposure to radiation using either beta blockers or non-dihydropyridine calcium channel blockers. According to North American Society for Cardiovascular Imaging (NASCI) recommendation in 2016, oral beta blocker prior to CCTA in patient with HR > 60 bpm is the preferred intervention. The recommended oral beta blocker usually is metoprolol 50-100 mg 1 hour prior to CCTA. The dosage of metoprolol must not exceed 400 mg/day. However, there are populations that are contraindicated or need to avoid beta blockers, such as uncontrolled obstructive airway disease, patient with baseline SBP < 100 mmHg, etc. Also, data in many clinical trials suggested that even high dose beta blockers can't controlled HR to target prior to CCTA in some patients. These pieces of information lead to alternative drugs to control HR prior to CCTA.

In previous clinical trials, the effective of non-dihydropyridine calcium channel blockers to control HR prior to CCTA compare to beta blockers had unclear results. In one study, Intravenous (IV) diltiazem is as effective in HR lowering to target to less than 60 bpm as IV metoprolol. Another study expressed inferior result of oral verapamil 1 hour before CCTA compared to oral metoprolol. However, there was heterogeneity in population of metoprolol and verapamil groups. According to FDA, immediate release (IR) diltiazem has onset of action faster than verapamil IR at 30 & 60-120 min., respectively. Initial dose of diltiazem in patients with chronic stable coronary artery disease and supraventricular tachycardia is at 30 - 60 mg oral every 6 hour and not exceed 360 mg/day.

Another agent that started to gain more evidence in HR control is ivabradine. Ivabradine has high selective and inhibitive property to If current channel which related to sinus node pace maker activity. Thus, other ion current channel normally doesn't get involved and doesn't have direct other cardiovascular effect. From meta-analysis, patients received ivabradine significantly achieving target HR to at least 65 bpm more than beta blockers group prior to CCTA (OR 5.02; 95% CI 3.16- 7.98, p < 0.00001, I 2 = 20%). In current recommendation, dosage of ivabradine shouldn't exceed 15 mg per day in patients with heart failure and chronic stable coronary artery disease. However, ivabradine has contraindication in patient with atrial fibrillation and/or sinus node disease, which require other agent to achieve target HR prior to CCTA. In current situation, there is no clinical trial to compare effect of beta blocker, non-dihydropyridine calcium channel blocker and Ivabradine in HR reduction to achieve target prior to CCTA.

The aim of this study is to compare percentage of patients achieving target HR < 60 bpm medication prior to CCTA by using oral beta blockers, non-dihydropyridine calcium channel blocker and ivabradine for HR lowering. Our study is double-blinded randomized controlled trial using Metoprolol immediate release as representative of beta blockers for controlled group, Diltiazem immediate release as representative of non-dihydropyridine calcium channel blocker and ivabradine. We blinded both investigators and patients using encapsulated drugs distribute from Siriraj's dispensary and randomly assign to our patients. The secondary objective of this study is to compare side effects, time to achieve target HR & CCTA image quality using 5 point grade scale and modified 15-segment American College of Cardiology and American Heart Association (AHA) between oral Metoprolol immediate, Diltiazem immediate release and ivabradine.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 year-old
2. Received Coronary CT angiography at Siriraj Hospital to evaluate diagnosis of coronary artery disease or risk stratification of coronary artery disease
3. Normal sinus rhythm with baseline HR > 60 bpm which cardiac imaging specialist suggest using HR lowering intervention

Exclusion Criteria:

1. Atrial fibrillation
2. Previous pacemaker implantation
3. II- and III-degree atrio-ventricular-block
4. NHYA class III - IV
5. Documented LVEF < 40%
6. Contraindication for CCTA: Impaired renal function (serum creatinine > 1.5 mg/dl), known allergy to iodinated contrast media, pregnancy, thyroid disease
7. Blood pressure < 100/70 mmHg
8. Uncontrolled asthma and/or chronic obstructive pulmonary disease (defined as GOLD stage D) and/or uncontrolled reactive airway disease
9. Current medication which cause severe interaction with calcium channel blocker, beta blocker and/or Ivabradine
10. Known allergy to calcium channel blocker, beta blocker and/or Ivabradine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent of patient achieving target heart rate (HR) | 3 hours
  To compare percentage of patient in achieving adequate HR control (defined as target HR of 60 bpm) among oral Ivabradine, metoprolol and diltiazem during CCTA

SECONDARY OUTCOMES:
Side effects | 3 hours
  To compare side effects between oral Ivabradine, metoprolol and diltiazem during CCTA
Time to achieve target HR | 3 hours
  To compare time to achieve target HR of less than 60 bpm
Image quality | 1 week
  To compare image quality using 5 point grade scale and modified 15-segment American College of Cardiology and American Heart Association (AHA)

CONTACTS AND LOCATIONS:
Overall Officials: Prichapol Thantassanee, M.D., Principal Investigator — Department of Internal Medicine, Faculty of Medicine, Siriraj Hospital Mahidol University
Locations (1):
- Department of Internal Medicine, Faculty of Medicine, Siriraj Hospital Mahidol University, Bangkok, Bangkoknoi, Thailand

REFERENCES:
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Mollet NR, Cademartiri F, van Mieghem CA, Runza G, McFadden EP, Baks T, Serruys PW, Krestin GP, de Feyter PJ. High-resolution spiral computed tomography coronary angiography in patients referred for diagnostic conventional coronary angiography. Circulation. 2005 Oct 11;112(15):2318-23. doi: 10.1161/CIRCULATIONAHA.105.533471. Epub 2005 Oct 3. PMID 16203914
- [Background] Raff GL, Gallagher MJ, O'Neill WW, Goldstein JA. Diagnostic accuracy of noninvasive coronary angiography using 64-slice spiral computed tomography. J Am Coll Cardiol. 2005 Aug 2;46(3):552-7. doi: 10.1016/j.jacc.2005.05.056. PMID 16053973
- [Background] Pugliese F, Mollet NR, Runza G, van Mieghem C, Meijboom WB, Malagutti P, Baks T, Krestin GP, deFeyter PJ, Cademartiri F. Diagnostic accuracy of non-invasive 64-slice CT coronary angiography in patients with stable angina pectoris. Eur Radiol. 2006 Mar;16(3):575-82. doi: 10.1007/s00330-005-0041-0. Epub 2005 Nov 16. PMID 16292649
- [Background] Giesler T, Baum U, Ropers D, Ulzheimer S, Wenkel E, Mennicke M, Bautz W, Kalender WA, Daniel WG, Achenbach S. Noninvasive visualization of coronary arteries using contrast-enhanced multidetector CT: influence of heart rate on image quality and stenosis detection. AJR Am J Roentgenol. 2002 Oct;179(4):911-6. doi: 10.2214/ajr.179.4.1790911. PMID 12239036
- [Background] Abbara S, Arbab-Zadeh A, Callister TQ, Desai MY, Mamuya W, Thomson L, Weigold WG. SCCT guidelines for performance of coronary computed tomographic angiography: a report of the Society of Cardiovascular Computed Tomography Guidelines Committee. J Cardiovasc Comput Tomogr. 2009 May-Jun;3(3):190-204. doi: 10.1016/j.jcct.2009.03.004. Epub 2009 Mar 31. No abstract available. PMID 19409872
- [Background] Qiu S, Shi S, Ping H, Zhou S, Wang H, Yang B. Efficacy of Ivabradine versus beta-Blockers for Heart Rate Reduction during Computed Tomography Coronary Angiography: A Meta-Analysis of Randomized Controlled Trials. Cardiology. 2016;135(3):133-140. doi: 10.1159/000447236. Epub 2016 Jun 22. PMID 27328446
- [Background] Maffei E, Palumbo AA, Martini C, Tedeschi C, Tarantini G, Seitun S, Ruffini L, Aldrovandi A, Weustink AC, Meijboom WB, Mollet NR, Krestin GP, de Feyter PJ, Cademartiri F. "In-house" pharmacological management for computed tomography coronary angiography: heart rate reduction, timing and safety of different drugs used during patient preparation. Eur Radiol. 2009 Dec;19(12):2931-40. doi: 10.1007/s00330-009-1509-0. PMID 19597820
- [Background] Degertekin M, Gemici G, Kaya Z, Bayrak F, Guneysu T, Sevinc D, Mutlu B, Aytaclar S. Safety and efficacy of patient preparation with intravenous esmolol before 64-slice computed tomography coronary angiography. Coron Artery Dis. 2008 Feb;19(1):33-6. doi: 10.1097/MCA.0b013e3282f27c20. PMID 18281813
- [Background] Shapiro MD, Pena AJ, Nichols JH, Worrell S, Bamberg F, Dannemann N, Abbara S, Cury RC, Brady TJ, Hoffmann U. Efficacy of pre-scan beta-blockade and impact of heart rate on image quality in patients undergoing coronary multidetector computed tomography angiography. Eur J Radiol. 2008 Apr;66(1):37-41. doi: 10.1016/j.ejrad.2007.05.006. Epub 2007 Jun 22. PMID 17587526
- [Background] Rochitte CE, Azevedo GS, Shiozaki AA, Azevedo CF, Kalil Filho R. Diltiazem as an alternative to beta-blocker in coronary artery computed tomography angiography. Arq Bras Cardiol. 2012 Aug;99(2):706-13. doi: 10.1590/s0066-782x2012005000059. Epub 2012 Jun 26. English, Portuguese. PMID 22735866
- [Background] Roberts WT, Wright AR, Timmis JB, Timmis AD. Safety and efficacy of a rate control protocol for cardiac CT. Br J Radiol. 2009 Apr;82(976):267-71. doi: 10.1259/bjr/24574758. Epub 2008 Dec 19. PMID 19098083
- [Background] Bois P, Bescond J, Renaudon B, Lenfant J. Mode of action of bradycardic agent, S 16257, on ionic currents of rabbit sinoatrial node cells. Br J Pharmacol. 1996 Jun;118(4):1051-7. doi: 10.1111/j.1476-5381.1996.tb15505.x. PMID 8799581
- [Background] DiFrancesco D, Camm JA. Heart rate lowering by specific and selective I(f) current inhibition with ivabradine: a new therapeutic perspective in cardiovascular disease. Drugs. 2004;64(16):1757-65. doi: 10.2165/00003495-200464160-00003. PMID 15301560
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Swedberg K, Komajda M, Bohm M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L; SHIFT Investigators. Ivabradine and outcomes in chronic heart failure (SHIFT): a randomised placebo-controlled study. Lancet. 2010 Sep 11;376(9744):875-85. doi: 10.1016/S0140-6736(10)61198-1. PMID 20801500
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Fox K, Ford I, Steg PG, Tendera M, Robertson M, Ferrari R; BEAUTIFUL Investigators. Relationship between ivabradine treatment and cardiovascular outcomes in patients with stable coronary artery disease and left ventricular systolic dysfunction with limiting angina: a subgroup analysis of the randomized, controlled BEAUTIFUL trial. Eur Heart J. 2009 Oct;30(19):2337-45. doi: 10.1093/eurheartj/ehp358. Epub 2009 Aug 31. PMID 19720635
- [Background] Fox K, Ford I, Steg PG, Tendera M, Ferrari R; BEAUTIFUL Investigators. Ivabradine for patients with stable coronary artery disease and left-ventricular systolic dysfunction (BEAUTIFUL): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Sep 6;372(9641):807-16. doi: 10.1016/S0140-6736(08)61170-8. Epub 2008 Aug 29. PMID 18757088
- [Background] Fox K, Ford I, Steg PG, Tardif JC, Tendera M, Ferrari R; SIGNIFY Investigators. Ivabradine in stable coronary artery disease without clinical heart failure. N Engl J Med. 2014 Sep 18;371(12):1091-9. doi: 10.1056/NEJMoa1406430. Epub 2014 Aug 31. PMID 25176136
- [Background] Pichler P, Pichler-Cetin E, Vertesich M, Mendel H, Sochor H, Dock W, Syeda B. Ivabradine versus metoprolol for heart rate reduction before coronary computed tomography angiography. Am J Cardiol. 2012 Jan 15;109(2):169-73. doi: 10.1016/j.amjcard.2011.08.025. Epub 2011 Oct 18. PMID 22011557